CLINICAL TRIAL: NCT04581551
Title: Reliability and Validity Study to Assess the Test-retest and Intra-rater Reliability of SWE in Shoulder Muscles in Persons After Stroke.
Brief Title: Reliability and Validity Study for SWE of Shoulder Muscles in Persons After Stroke.
Acronym: SWE_stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: B6702020000601
Record Dates: First submitted 2020-09-09; First posted 2020-10-09 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-06

CONDITIONS: Stroke
Keywords: Stroke; Shear wave elastography; Shoulder muscles; Shoulder pain
MeSH Terms: conditions — Stroke; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke group (Experimental): SWE for 6 shoulder muscles will be performed by 2 assessors in randomised order.
  * m. supraspinatus
  * m. infraspinatus
  * m. rhomboideus major
  * m. deltoideus
  * m. pectoralis major
  * m. pectoralis minor
  Interventions: Procedure: SWE assessor 1; Procedure: SWE assessor 2; Procedure: Stretch intervention; Procedure: No stretch intervention
- Healthy controls (Active Comparator): SWE for 6 shoulder muscles will be performed by 1 assessors.
  * m. supraspinatus
  * m. infraspinatus
  * m. rhomboideus major
  * m. deltoideus
  * m. pectoralis major
  * m. pectoralis minor
  Interventions: Procedure: SWE assessor 1

INTERVENTIONS:
Procedure: SWE assessor 1 — SWE for 6 shoulder muscles will be performed.
  * m. supraspinatus
  * m. infraspinatus
  * m. rhomboideus major
  * m. deltoideus
  * m. pectoralis major
  * m. pectoralis minor
Procedure: SWE assessor 2 — SWE for 6 shoulder muscles will be performed.
  * m. supraspinatus
  * m. infraspinatus
  * m. rhomboideus major
  * m. deltoideus
  * m. pectoralis major
  * m. pectoralis minor
  Arms: Stroke group
Procedure: Stretch intervention — Transversal stretch of pectoralis major muscle on the hemiplegic side.
  Arms: Stroke group
Procedure: No stretch intervention — Passive mobilisation of the hemiplegic hand.
  Arms: Stroke group

SUMMARY:
This study aims

1. To examine the reliability of SWE assessment in the shoulder muscles of persons after a stroke.
2. To assess if differentiation can be made between the hemiplegic (HP) and non-hemiplegic (NHP) side and between stroke patients and matched healthy volunteers (discriminative validity).
3. To assess if an immediate effect on the pectoralis major and minor can be measured after applying transversal stretch technique to the pectoralis major muscles (response validity).

DETAILED DESCRIPTION:
Stroke patients will be assessed on 2 days with an interval of 3 days (Friday - Monday).

Day 1 (Friday): shear wave velocity (SWV) will be assessed by 2 assessors in randomised order. Each assessor will evaluate SWV of 6 shoulder muscles (m. supraspinatus, m. infraspinatus, m. rhomboid major, m. deltoideus, m. pectoralis major, m. pectoralis minor).

At the end of the assessment secondary outcome measures will be assessed.

Day 2 (Monday): SWV will be reassessed by assessor 1 to measure test-retest reliability.

Position of the patient will be changed. SWV of the pectoralis major and minor muscle will be reassessed.

Assessor 2 will perform a transversal stretch of the m. pectoralis major or a passive mobilisation of the hand at the hemiplegic arm of the stroke patients. Assessor 1 will reassess the SWV of the pectoralis major and minor muscle to assess if there is an immediate effect of the intervention. Assessor 1 will be blinded for the intervention.

Healthy controls (matched for age, gender and BMI):

Only one test day to assess SWV of 6 shoulder muscles. Secondary outcome measures will be assessed after SWE assessment.

ELIGIBILITY:
Stroke group

Inclusion:

* Stroke patients in the subacute phase after stroke (< 6 months post stroke)
* Able to sit independently with support of the back, but without support of the arms
* With upper-limb (UL) impairment: i.e. no maximum score (36) on the shoulder elbow part of the Fugl-Meyer UL (FM UL)

Exclusion Criteria:

* Other neurologic disorders
* Shoulder or neck surgery before stroke onset
* Arthroscopic surgery in the last year before stroke onset.
* Shoulder or neck pain in the last year before stroke onset.
* Severe cognitive or language deficits that inhibit the participants of understanding simple commands or providing valuable information regarding the outcome measures - measured with the Ability Q.
* Participants who are not able to maintain the test position.
* Pregnancy

Healthy controls can participate if they

* Have not suffered a stroke or other neurological disorders
* Did not have surgery at the shoulder and/or neck
* Did not have arthroscopic surgery in the last year before stroke
* If they do not suffer any shoulder or neck pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
SWV m. supraspinatus | Single point of assessment on day 1 (test)
  Shear wave velocity of the m. supraspinatus
SWV m. supraspinatus | Single point of assessment on day 2 (retest)
  Shear wave velocity of the m. supraspinatus
SWV m. infraspinatus | Single point of assessment on day 1 (test)
  Shear wave velocity of the m. infraspinatus
SWV m. infraspinatus | Single point of assessment on day 2 (retest)
  Shear wave velocity of the m. infraspinatus
SWV m. rhomboideus major | Single point of assessment on day 1 (test)
  Shear wave velocity of the m. rhomboideus major
SWV m. rhomboideus major | Single point of assessment on day 2 (retest)
  Shear wave velocity of the m. rhomboideus major
SWV m. deltoideus | Single point of assessment on day 1 (test)
  Shear wave velocity of the m. deltoideus
SWV m. deltoideus | Single point of assessment on day 2 (retest)
  Shear wave velocity of the m. deltoideus
SWV m. pectoralis major | Single point of assessment on day 1 (test)
  Shear wave velocity of the m. pectoralis major
SWV m. pectoralis major | Single point of assessment on day 2 (retest)
  Shear wave velocity of the m. pectoralis major
SWV m. pectoralis minor | Single point of assessment on day 1 (test)
  Shear wave velocity of the m. pectoralis minor
SWV m. pectoralis minor | Single point of assessment on day 2 (retest)
  Shear wave velocity of the m. pectoralis minor

SECONDARY OUTCOMES:
Demographic variables | Baseline assessment day 1
  Age, gender, weight, height, dominance, date of birth, stroke date, type of stroke, side of paresis
Passive range of motion of shoulder | Baseline assessment day 1
  Goniometric measurement of shoulder flexion, abduction, external rotation, internal rotation (degrees)
Spasticity shoulder muscles | Assessment day 1
  Modified Ashworth Scale (minimum 0 - maximum 4, higher score is more spasticity = worse outcome) of shoulder flexors, extensors, internal rotators, external rotators, adductors, abductors
Shoulder subluxation - ultrasound measurement | Assessment day 1
  Acromiohumeral distance of the hemiplegic and non-hemiplegic shoulder subtracted
Fugl-Meyer assessment upper limb section | Assessment day 1
  Active recovery of the upper limb motor function
Subjective feeling of shoulder stiffness | Assessment day 1
  Question to the patients about how stiff the shoulder feels
Sports before stroke | Assessment day 1
  Question if stroke patients performed sports before stroke and which sports they performed before stroke

OTHER OUTCOMES:
Subcutaneous tissue thickness | Single point of assessment on day 1
  Measurement de thickness of the subcutaneous layer on the ultrasound image of the m. pectoralis major to compare the stroke group and healthy control group.

CONTACTS AND LOCATIONS:
Overall Officials: Annelies Maenhout, Prof, Principal Investigator — University Ghent; Kristine Oostra, Prof, Principal Investigator — University Hospital, Ghent; Dirk Cambier, Prof, Principal Investigator — University Ghent
Locations (2):
- Belgium (2):
  - Ghent University Hospital, Ghent
  - Ghent University, Ghent

IPD SHARING:
Plan to Share IPD: No